CLINICAL TRIAL: NCT02038972
Title: Safety of Autologous Stem Cell Infusion for Children With Acquired Hearing Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: James Baumgartner, MD (Other)
Collaborators: CBR Systems, Inc. (Other)
Responsible Party: Sponsor-Investigator, James Baumgartner, MD, Primary Investigator, AdventHealth
Organization: AdventHealth (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 434269
Record Dates: First submitted 2014-01-08; First posted 2014-01-17 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2017-08

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Autologous Stem Cells (Experimental): A single dose of intravenously administered autologous hUCB will be done. The minimum acceptable dose will be 6x10 6th mononuclear cells/kilogram body weight. The hUCB reanimation, cell processing and product infusion will occur at Florida Hospital for Children and the Florida Hospital Center for Cellular Therapy.
  Interventions: Genetic: Autologous Stem Cells

INTERVENTIONS:
Genetic: Autologous Stem Cells — The subjects autologous stem cells banked at Cord Blood Registry will be infused intravenously by gravity.
  Other Names: Cell based therapy

SUMMARY:
To determine if autologous human umbilical cord blood infusion in children with acquired hearing loss is safe, feasible, improves inner ear function, audition and language development.

DETAILED DESCRIPTION:
There is currently no treatment available to repair/reverse acquired sensorineural hearing loss. Recent experiments using human umbilical cord blood treatment of a mouse and guinea pig models have demonstrated hair cell re-growth following acquired sensorineural loss as well as partial restoration of ABR. Autologous human umbilical cord blood therapy, which has been used for over twenty years, has an excellent safety record. This study will determine if autologous human umbilical cord blood infusion in children with hearing loss is safe and feasible, improves inner ear function, audition, and language development. The patients umbilical cord stem cells collected at birth and stored at Cord Blood Registry will be used for infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a sensorineural hearing loss

   * Unilateral or bilateral in configuration
   * Symmetrical or asymmetrical configuration
   * Sudden or progressive in presentation
   * Moderate to profound in degree (40-90 Decibels (dB) in at least one ear
2. Normally shaped cochlea, as determined by MRI
3. The loss must be considered:

   * Acquired
   * Unknown with a negative genetic test.
4. Fitted for hearing aids no later than six months post detection of loss.
5. Enrollment in a parent/child intervention program
6. Age 6 weeks - 6 years old at time of infusion with less than 18 months of hearing loss at the time of cord blood infusion.
7. Ability of the child and caregiver to travel to Orlando, and stay for at least 4 days, and to return for all follow-up visits.

Exclusion Criteria

1. Inability to obtain all pertinent medical records:

   * (pertinent physician notes, speech language pathology notes, laboratory findings, test results and imaging studies-must be sent to the research team at least prior to the subject arriving at the study location for preliminary screening and eligibility assessment, preferably14 days before the scheduled hUBC treatment.)
2. Known history of:

   * Recently treated infection less than 2 weeks before infusion.
   * Renal disease of altered renal function as defined by serum creatinine > 1.5 mg/dl at admission.
   * Hepatic disease or altered liver function as defined by SGPT > 150 U/L, and or T. Bilirubin > 1.3 mg/dL
   * Malignancy
   * Immunosuppression as defined by WBC < 3,000 at admission
   * Human Immunodeficiency Virus (HIV)
   * Hepatitis B
   * Hepatitis C
   * Evidence of an extensive stroke (> 100ml lesion)
   * Pneumonia, or chronic lung disease requiring oxygen
   * Genetic syndromic sensorineural hearing loss
3. hUBC sample contamination
4. Banked cord cells totaling less than 6x106 mononuclear cells/kilogram body weight.
5. Evidence of the following maternal infections during the pregnancy (Hepatitis A, Hepatitis B, Hepatitis C, HIV 1, HIV 2, Human T-lymphotropic Virus (HTLV) 1, HTLV 2 (CMV and Syphilis can be included in the study)
6. participation in a concurrent intervention study
7. Unwillingness or inability to stay for 4 days following hUBC infusion (should problems arise following the infusion) and to return for the one month, six month and one year follow-up visits.
8. Presence of a cochlear implantation device
9. Evidence of a genetic syndrome
10. Evidence of conductive hearing loss
11. Documented recurrent middle ear infections which are frequent (>5 per year)
12. Otitis media at the time of examination
13. Sensorineural loss is mild
14. Over 18 months from identification of hearing loss at time of infusion

Ages: 6 Weeks to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12-11 (Actual); Study Completion 2017-01-10 (Actual)

PRIMARY OUTCOMES:
Safety of Autologous Stem Cell Infusion | 1 year
  To determine if autologous human umbilical cord blood (hUBC) infusion in children with hearing loss is safe and feasible. Infusion related toxicity as measured by:
  i. hemodynamic instability: An adverse event will be defined as a sustained (> 10 minutes) >20% decrease in MAP.
  ii. acute lung injury: Chest X-ray will be done at baseline and at 1 day post infusion to assess for polymorphonuclear infiltrates iii. hepatic injury/toxicity: Hepatic panel will be performed at baseline and 1 day post infusion. Injury is defined as acute elevation of the AST/ALT hepatic enzymes > 900 U/dl in the first 24 hours post infusion iv. renal injury/insufficiency: CMP will be performed at baseline and 1 day after infusion v. exacerbation of neurological status: defined as a change in Glasgow Coma Scale, pupillary size/reactivity, motor/sensory evaluation of extremities, and seizure activity from infusion to discharge.

SECONDARY OUTCOMES:
Inner Ear Function, Audition, and Language Development | 1 year
  To determine if autologous hUBC transplantation in children with hearing loss improves inner ear function, audition and language development.

CONTACTS AND LOCATIONS:
Overall Officials: James Baumgartner, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided